CLINICAL TRIAL: NCT02474953
Title: A Randomized, Double-blind, Crossover Study to Compare the Pharmacokinetic Profile of a Proprietary Curcumin Formulation to a Comparator Curcumin Product
Brief Title: A Study to Compare the Pharmacokinetic Profile of a Proprietary Curcumin Forumulation to a Comparator Curcumin Product
Acronym: 15PCHB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Boston Biopharm, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 15PCHB
Record Dates: First submitted 2015-06-10; First posted 2015-06-18 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Curcumin; Pharmacokinetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dosing Sequence 1 (Experimental): Proprietary Curcumin Formulation administered first, Unformulated Comparator Curcumin Product administered second
  Interventions: Dietary Supplement: Proprietary Curcumin Formulation; Dietary Supplement: Unformulated Comparator Curcumin Product
- Dosing Sequence 2 (Experimental): Unformulated Comparator Curcumin Product administered first, Proprietary Curcumin Formulation administered second
  Interventions: Dietary Supplement: Proprietary Curcumin Formulation; Dietary Supplement: Unformulated Comparator Curcumin Product

INTERVENTIONS:
Dietary Supplement: Proprietary Curcumin Formulation
Dietary Supplement: Unformulated Comparator Curcumin Product

SUMMARY:
This study is investigating the pharmacokinetic profile (i.e. the way the product is processed by the body) of a proprietary curcumin formulation compared to an unformulated curcumin product. Subjects will take a single dose of either the proprietary formulation or comparator product and the blood levels of curcumin and curcumin metabolites will be measured over a period of 48 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females 18-45 years of age
2. If female, subject is not of child bearing potential, which is defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) OR

   Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Non-hormonal intrauterine devices
   * Vasectomy of partner
3. BMI 18-29.9 kg/m2 (±1 kg/m2)
4. Healthy as determined by laboratory results and medical history
5. Agrees to maintain current level of physical activity throughout the study
6. Agree to avoid using black or white pepper, turmeric, curcumin or curry in the preparation of food for 7 days prior to randomization and throughout the study period.
7. Agree to avoid Indian and Thai cuisines for the period of the study
8. Agree to avoid food with yellow dye #E100
9. Agrees to avoid alcohol, caffeine 12 hours and grapefruit and grapefruit juice 48 hours prior to baseline and each subsequent clinic visit
10. Agrees to consume only low polyphenols in the diet (nutritionists will counsel on high polyphenol fruits, vegetables to avoid, wine, beer, supplements, herbal extracts, and whole-grain based foods) 3 days prior to baseline and on test days (meal options and lists of foods to avoid will be provided to subjects by nutritionists)
11. Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. BMI ≥ 30 kg/m2
2. Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial.
3. Unstable medical conditions as determined by the Qualified Investigator
4. Use of natural health products containing turmeric or curcumin within 7 days prior to randomization and during the course of the study
5. Use of St Johns Wort 3 weeks prior to baseline and during the study
6. Subjects who are smokers
7. Subjects with current or history of gastrointestinal problems or disease
8. Metabolic, endocrine, or chronic diseases
9. Immunocompromised individuals such as subjects that have undergone organ transplantation or subjects diagnosed with human immunodeficiency virus (HIV)
10. Clinically significant abnormal lab results at screening (e.g. AST and/or ALT > 2 x ULN, and/or bilirubin > 2 x ULN) will be assessed by the Qualified Investigator
11. Subjects who have planned surgery during the course of the trial
12. History of or current diagnosis of any cancer (except for successfully treated basal cell carcinoma) diagnosed less than 5 years prior to screening. Subjects with cancer in full remission more than 5 years of diagnosis are acceptable.
13. History of gallbladder issues, hyperacidity, gastric/duodenal ulcers.
14. Prior use of prescription H2 blocker, proton pump inhibitor or blood sugar-lowering agents
15. Use of blood pressure medication
16. Subjects on restrictive dietary regimens
17. Blood donation in the last 2 months
18. History of blood/bleeding disorders or taking prescription blood thinners or anti-platelet therapy
19. Alcohol abuse (>2 standard alcoholic drinks per day) or drug abuse within the past 6 months
20. Use of medical marijuana
21. Clinically significant abnormal laboratory results at screening
22. Participation in a clinical research trial within 30 days prior to randomization
23. Allergy or sensitivity to study supplement ingredients or to any food or beverage provided during the study
24. Individuals who are cognitively impaired and/or who are unable to give informed consent
25. Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Curcumin AUC | Time 0 to 48 hours
  Area Under the Curve
Curcumin Cmax | Time 0 to 48 hours
  Maximum Concentration
Curcumin Tmax | Time 0 to 48 hours
  Time until maximum concentration

OTHER OUTCOMES:
Incidence of adverse events | Time 0 to 48 hours
Changes in blood CBC levels | Time 0 to 48 hours
Changes in blood electrolyte levels | Time 0 to 48 hours
Changes in blood creatinine levels | Time 0 to 48 hours
Changes in blood AST levels | Time 0 to 48 hours
Changes in blood ALT levels | Time 0 to 48 hours
Changes in blood GGT levels | Time 0 to 48 hours
Changes in blood bilirubin levels | Time 0 to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada